CLINICAL TRIAL: NCT03841955
Title: A Prospective, Multicentre, Randomized, Open, Parallel Controlled Clinical Trial for Evaluating the Safety and Effectiveness of CATHTONG™ II PICC
Brief Title: Safety and Effectiveness of CATHTONG™ II PICC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PICC-2017-1016
Record Dates: First submitted 2019-01-23; First posted 2019-02-15 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2020-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Catheterization, Peripheral

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Peripheral implantation of central venous catheters and accessories with high pressure tolerance
  Interventions: Device: PICC with high pressure tolerance
- Control group (Experimental): Peripheral intubation of central venous catheter
  Interventions: Device: rontine central venous catheter

INTERVENTIONS:
Device: PICC with high pressure tolerance — Subjects signed informed consent, meet the inclusion criteria and did not meet the exclusion criteria, and were randomly admitted to the experimental group and given the intervention.
  Other Names: Peripheral intubation of central venous catheter
  Arms: Experimental group
Device: rontine central venous catheter — Subjects signed informed consent, meet the inclusion criteria and did not meet the exclusion criteria, and were randomly admitted to the control group and given the intervention.
  Arms: Control group

SUMMARY:
This clinical trial is a prospective, multi-centre, open, parallel and comparative non-inferior trial design.

DETAILED DESCRIPTION:
Four clinical trial institutions that meet the national qualification are selected as clinical research centers. After informed consent of the subjects and meeting the selection criteria, the subjects will be included in this clinical study. After the follow-up, all the data were sorted out and analyzed. Finally, the data of the two groups were compared to prove whether the high-pressure-resistant peripherally inserted central venous catheter developed by L&Z US, Inc. was not inferior to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects volunteered to participate in the trial and signed the informed consent.
* Age 18 years old, 80 years old; gender is not limited;
* Suitable for patients who need central venous catheterization via peripheral venipuncture (life expectancy is more than 6 months): need medium-term and long-term infusion or intravenous drug therapy; need multi-chamber infusion of multiple drugs at the same time; need infusion of irritating, corrosive or hyperosmotic drugs; hyperbaric angiography or central venous pressure monitoring function;
* Patients who need to be maintained in the investigator's hospital after PICC catheterization;
* Ability to communicate well with researchers and comply with test requirements.

Exclusion Criteria:

* Local infection of puncture vein or occlusion or serious lesion of blood vessel at puncture place;
* Patients with known or suspected allergies to polyurethane;
* Pre-intubation site includes trauma history, vascular surgery history, thrombosis history, radiotherapy history, bilateral breast cancer surgery affected upper limbs, superior vena cava compression syndrome, etc.
* The prothrombin time was 6 seconds longer than the normal value and the activated partial thromboplastin time was 2.5 times longer than the normal value.
* Pregnancy and lactation women;
* The subjects had a history of difficulty in catheterization.
* Patients with pacemaker implantation in vivo;
* Researchers do not consider it appropriate to participate in this clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Successful rate of one-time catheterization | Day 1
  Subcutaneous detection of blood vessel movements less than three times, and finally completed catheterization and confirmed that the end of the catheter in the pre-positioning proportion of the total number of patients (catheterization success refers to the chest X-ray and other fluoroscopy means to confirm that the end of the catheter is located in the middle and lower segment of superior vena cava).

SECONDARY OUTCOMES:
Operating time | Day 1
  The time between the beginning of disinfection of the patient's skin and the fixing of transparent dressing is in minutes.
success rate of one puncture. | Day 1
  Success of one puncture refers to entering the target vein only once. If the puncture needle failed to penetrate the vein once and retreated to the subcutaneous area, then exploratory puncture was the second puncture.
The incidence of adverse events | about three months
  Record the adverse events in the test, determine whether they are related to the test product, and calculate the incidence of adverse events/reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Jin jingfen, Master, Principal Investigator — The second affiliated hosital of medical college of zhejiang university
Locations (4):
- China (4):
  - Affiliated Cancer Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial Tongde Hospital, Hangzhou, Zhejiang
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided